CLINICAL TRIAL: NCT05758623
Title: Mg-containing Biodegradable Polymer Bone Repair Material
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Zhongke Jingcheng Medical Technology Co., Ltd (Other)
Collaborators: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P_204970118082038
Record Dates: First submitted 2023-02-13; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Bone Deformity
MeSH Terms: interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium containing biodegradable polymer bone repair material (Placebo Comparator): The experimental group was treated with magnesium containing biodegradable polymer bone repair material produced by Shenzhen Zhongke Jingcheng Medical Technology Co., Ltd.
  Interventions: Device: Device
- β- Tricalcium phosphate bioceramics (Placebo Comparator): Control group application β- Tricalcium phosphate bioceramics for treatment.
  Interventions: Device: Device

INTERVENTIONS:
Device: Device — The experimental group was treated with magnesium containing biodegradable polymer bone repair material produced by Shenzhen Zhongke Jingcheng Medical Technology Co., Ltd. Control group application β- Tricalcium phosphate bioceramics for treatment.

SUMMARY:
The subjects of this study are patients with non-load-bearing bone defects of the extremities who need bone grafting surgery. The patients was treated with bone graft using magnesium containing biodegradable polymer bone repair material produced by Shenzhen Zhongke Jingcheng Medical Technology Co., Ltd.. Three follow-up visits were performed at the 12th, 24th and 36th weeks after bone grafting, the clinical role for bone will be assessed.

DETAILED DESCRIPTION:
The subjects of this study are patients with non-load-bearing bone defects of the extremities who need bone grafting surgery. The subjects were randomly divided into experimental group and control group. The experimental group was treated with bone graft using magnesium containing biodegradable polymer bone repair material produced by Shenzhen Zhongke Jingcheng Medical Technology Co., Ltd., while the control group was treated with bone graft β- Tricalcium phosphate bioceramics were used for bone transplantation. Three follow-up visits were performed at the 12th, 24th and 36th weeks after bone grafting. It is estimated that 176 cases will be recruited in total, and 135 cases have been recruited since April 2021. This product can be degraded and absorbed in vivo, and it can promote the formation of new bone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 75 years old, regardless of gender;
2. Bone defect exists in one of the following anatomical positions, and bone grafting is required:

   Upper limb bones: humerus, ulna, radius, metacarpus, carpus, phalanges;

   Lower limb bones: femur, tibia, fibula, calcaneus, navicular bone, wedge bone, cuboid bone, metatarsal bone, talus and phalanges;
3. The maximum diameter of the expected or actual three-dimensional bone defect is ≥ 0.5cm and ≤ 6cm, and the defect is only one;
4. The bone defect site is expected to be fixed with non-degradable internal fixation system during operation;
5. Subjects or their legal representatives can understand the purpose of the study and show sufficient compliance with the study protocol and sign the informed consent form.

Exclusion Criteria:

1. The blood glucose control is unstable and cannot meet the operation conditions;
2. Severe coagulation dysfunction (PT or APTT ≥ 2 times the upper limit of normal value);
3. History of arterial thrombosis attack (such as stroke, angina pectoris, acute myocardial infarction, etc.) or NYHA grade ≥ III within 3 months before enrollment;
4. Oral or injection of sedative and hypnotic drugs or non-steroidal anti-inflammatory drugs (except aspirin) every week within 3 months before enrollment;
5. He had received chemotherapy drugs or radiotherapy within 3 months before admission;
6. Cumulative oral or injection of corticosteroids or various growth factors for ≥ 14 days within 1 month before enrollment;
7. Suffering from systemic infection or uncontrollable local infection, serious soft tissue injury at the proposed operation site, serious vascular or nerve injury, malignant tumor, confirmed severe malnutrition or other important organ failure;
8. The limb to be operated on has osteofascial compartment syndrome;
9. Structural bone grafting is required;
10. Pregnant or lactating women;
11. Participate in clinical trials of other drugs or medical devices within one month before enrollment;
12. For the benefit of the subject, the researcher believes that it should not participate in other situations of this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Bone graft fusion rate | 24 weeks after standard operation
  When Mg-containing degradable polymer bone repair material is used to repair non-load-bearing bone defects of limbs, the main effective evaluation index is bone graft fusion rate at 24 weeks after operation

SECONDARY OUTCOMES:
to evaluate the bone graft fusion rate | 12 and 36 weeks after operation
  to evaluate the bone graft fusion rate at 12 and 36 weeks after operation
Improvement level of SF-36 scale and satisfaction of device operation | at 36 weeks after operation
  Improvement level of SF-36 scale and satisfaction of instrument operation at 36 weeks after operation

CONTACTS AND LOCATIONS:
Overall Officials: Yuxiao Lai, Professor, Principal Investigator — Ext:+86 755 86392581 Email:Yx.Lai@siat.ac.cn Shenzhen Institute of Advanced Technology, Chinese Academy of Sciences; Ling Qin, Professor, Study Director — Ext:+86-755-86392258 Email:lingqin@cuhk.edu.hk The Chinese University of Hong Kong
Locations (1):
- Shenzhen Zhongke Jingcheng Medical Technology Co., Ltd, Shenzhen, Guangdong, China